CLINICAL TRIAL: NCT05727722
Title: A Phase I Safety and Tolerability Dose Escalation Study of Micro-encapsulated Hepatocytes Intraperitoneal Transplantation Therapy for Adult Liver Failure Patients.
Brief Title: Micro-encapsulated Hepatocyte Intraperitoneal Transplantation in Liver Failure Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Institute of Biochemistry and Cell Biology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT02-ProliHH-I
Record Dates: First submitted 2022-11-23; First posted 2023-02-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Acute-On-Chronic Liver Failure; Chronic Liver Failure
Keywords: Acute-On-Chronic Liver Failure; Chronic Liver Failure; cell transplantation; hepatocyte transplantation; micro-encapsulate
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; End Stage Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Micro-encapsulated Hepatocyte Intraperitoneal Transplantation Cohort 1 (Experimental): Participants will each be administered the dosage of 0.15×10^9 for one time, with 60 days follow-up after the cell infusion.
  Interventions: Biological: a single course of micro-encapsulated hepatocytes intraperitoneal transplantation therapy
- Micro-encapsulated Hepatocyte Intraperitoneal Transplantation Cohort 2 (Experimental): Participants will each be administered the dosage of 0.5×10^9 for one time, with 60 days follow-up after the cell infusion.
  Interventions: Biological: a single course of micro-encapsulated hepatocytes intraperitoneal transplantation therapy
- Micro-encapsulated Hepatocyte Intraperitoneal Transplantation Cohort 3 (Experimental): Participants will each be administered the dosage of 1.5×10^9 for one time, with 60 days follow-up after the cell infusion.
  Interventions: Biological: a single course of micro-encapsulated hepatocytes intraperitoneal transplantation therapy
- Micro-encapsulated Hepatocyte Intraperitoneal Transplantation Cohort 4 (Experimental): Participants will each be administered the dosage of 4.5×10^9 for one time, with 60 days follow-up after the cell infusion.
  Interventions: Biological: a single course of micro-encapsulated hepatocytes intraperitoneal transplantation therapy

INTERVENTIONS:
Biological: a single course of micro-encapsulated hepatocytes intraperitoneal transplantation therapy — A single course will be divided into an "accelerated titration design" phase and a "3+3 design" phase to reduce the number of subjects exposed to potentially ineffective doses that may not benefit from treatment. The "accelerated titration design" phase starts at a starting dose of 0.15x10^9, moving to the "3+3 design" phase at the dose of 0.5x10^9. According to the semi-logarithmic incremental (10^0.5-fold) approach, the treatment dosage was set into four groups at a maximum dose of 4.5×10^9 (allowing for a ±20% difference between the actual dose and the planned dose, considering production specifics). The number or the incremental ratio of subsequent dose groups can be adjusted based on the evaluation of available data in the study, and intermediate doses can be explored.

SUMMARY:
This is a prospective single-center dose escalation study of the administration of the microencapsulated hepatocyte therapy in adult liver failure. The purpose of the study is to determine the maximum tolerated dose of microencapsulated hepatocytes in liver failure patients and its effectiveness in treating the disease. We previously generated proliferating human hepatocytes (ProliHH) through dedifferentiation of PHH and engineered them into encapsulated liver organoids (eLO), providing an unlimited cell source for hepatocyte transplantation.

DETAILED DESCRIPTION:
This study is a single-center unblinded single-arm study comprised of a dose escalation phase and a preliminary assessment of efficacy. Subjects who were diagnosed with liver failure (including chronic liver failure and acute-on-chronic liver failure) received 3 days' regular treatment with no beneficial effect and volunteered to participate in micro-encapsulated hepatocytes intraperitoneal transplantation therapy will be enrolled. Before the clinical research, the recruitment criteria and micro-encapsulated hepatocytes transplantation protocol will be confirmed. To minimize the number of patients receiving unbeneficial therapeutic dosage, the accelerated titration design and "3+3" design will be used to decide the dosage group. All micro-encapsulated hepatocytes transplantation patients will be monitored after 1, 3, 7, 14, 28, and 60 days after treatment for safety and primary efficacy analyses. The patients could still receive regular clinical treatment including liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

A. Chronic liver failure (CLF) group:

The progressive liver function decline or decompensation after liver cirrhosis:

1. Body weight>40kg;
2. Aged between 18 to 65 years old;
3. Serum Total bilirubin was higher than the normal range and lower than 10 times the upper limit of normal value (ULN);
4. With or without significantly decreased serum albumin value, lower than 35;
5. With or without significantly decreased platelet (PLT) value, prothrombin activity (PTA)≤40% (or international normalized ratio (INR)≥1.5), other reasons excluded;
6. With or without refractory ascites or portal hypertension;
7. With or without a stage I or II hepatic encephalopathy;
8. No obvious improvement after more than 3 days' regular clinical treatments.

OR B. Acute-on-chronic liver failure (ACLF) group:

With known or unknown basic liver diseases, subjects undergoing acute liver failure syndrome (clinical manifestations indicated as an early stage liver failure).

1. Body weight>40kg;
2. Aged between 18 to 65 years old;
3. With obvious fatigue, accompanied by other gastrointestinal symptoms such as anorexia, vomiting, and abdominal distension;
4. Complicated with ascites and/or hepatic encephalopathy within 4 weeks after being diagnosed;
5. Progressive aggravation of jaundice, total serum bilirubin≥85umol/L；
6. Coagulation disorders, INR>1.5 or PTA<40%;
7. No obvious improvement after more than 3 days' regular clinical treatments.

Exclusion Criteria:

1. With obvious brain edema, cerebral hernia, or indicated intracranial hemorrhage;
2. Diagnosed or suspected as primary or metastatic liver cancer;
3. With uncorrectable oxygenation index (PaO2/FiO2)<200;
4. With disseminated intravascular coagulation;
5. Active hemorrhage;
6. Uncontrollable infection, including ascites infection such as spontaneous bacterial peritonitis;
7. Uncorrectable decrease in PLT (<20×109/L);
8. HIV and/or SARS-CoV-Ⅱ positive;
9. Drug abuse within 1 year;
10. Systemic hemodynamic instability;
11. Combined with pregnancy or lactation;
12. Other situations excluded by clinician;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events | baseline to 60 days after cell transplantation therapy
  All adverse events are defined and graded following the National Cancer Institute-Common Terminology Criteria for Adverse Events V.5.0. Adverse events (AE), serious adverse events (SAE), and treatment emergent AEs (TEAE)
Maximum tolerated dose (MTD) | baseline to 60 days after cell transplantation therapy
  The maximum tolerated dose (MTD) is defined as the highest dose at which no more than 1 of at least 6 subjects developed dose-limiting toxicity (DLT). During the DLT observation period, another patient should be enrolled if one subject does not complete the DLT observation period due to withdrawal for reasons other than DLT.

SECONDARY OUTCOMES:
Model for end-stage liver disease (MELD) score system | baseline to 60 days after cell transplantation therapy
  Laboratory test results used to calculate the MELD score must be obtained at the same time point, and the results need to be obtained within 6 hours of the blood draw.
The survival rates compared with historical controls | the 60th day after cell transplantation therapy
  The life table method was used to calculate the survival rate of patients.
Serum antibodies against human leukocyte antigen (HLA) Class I and II | baseline to 60 days after cell transplantation therapy
  The serum antibodies against HLA Class I and II are used to for immunogenicity evaluation.
Incidence of Clinical improvement | baseline to 60 days after cell transplantation therapy
  diagnosed refer to Chapter 2.6.2.2 of Guidelines for the Diagnosis and Management of Liver Failure (2018, China).

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

REFERENCES:
- [Derived] Yang T, Zhu X, Long M, Hui L, Yuan X, Sun Z, Zhang L, Xia Q, Wan P. Phase I safety and tolerability dose escalation study of microencapsulated hepatocyte intraperitoneal transplantation therapy in adult patients with liver failure: a study protocol. BMJ Open. 2025 Apr 15;15(4):e087828. doi: 10.1136/bmjopen-2024-087828. PMID 40233953